CLINICAL TRIAL: NCT05193240
Title: Predictive Value of a Preliminary Swallowing Test Compared to Postoperative Nasofibroscopy to Identify Vocal Cord Paralysis After Pulmonary Resection
Acronym: SwaLO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/0419/HP
Record Dates: First submitted 2021-12-27; First posted 2022-01-14 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2021-12

CONDITIONS: Adults Patients Undergoing Major Lung Resection in the Context of Lung Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- preliminary swallowing test (Experimental): compared as nasofibroscopy and ultrasound examination of vocal cords
  Interventions: Diagnostic Test: preliminary swallowing test

INTERVENTIONS:
Diagnostic Test: preliminary swallowing test — Patients will be included before the surgery. During this inclusion visit, we will perform a preoperative swallowing test.
  Immediately after surgery (H2-H24 after extubation), we will perform a preliminary swallowing test, an ultrasound examination of the vocal cords and a nasofibroscopy to determine the mobility of the vocal cords. A physiotherapist will carry out the first two assessments. An ENT physician will perform the nasofibroscopy. The ENT physician performing the nasofibroscopy will not know the conclusions of the tests carried out by the physiotherapist immediately after the operation.
  At last, on day 4 after extubation, we will repeat the preliminary swallowing test and the ultrasound examination to measure the evolution of cord mobility.
  30 days after the surgery, we will realize a follow-up on medical file and mark the end of the research.
  Other Names: nasofibroscopy; ultrasound examination of the vocal cords

SUMMARY:
The literature describes recurrent nerve damage during thoracic surgery as a fairly complication (5 to 31% of patients). This nerve damage leads to paresis or paralysis of the ipsilateral vocal cord. This cord dysfunction no longer ensures the protective role of the airways during swallowing. This postoperative dysphagia is associated with complications such as aspiration pneumonia, the use of nasogastric tube feeding (adding difficulty to swallowing), delayed oral refeeding (risk of undernutrition, dehydration, decrease in the quality of life), and an increase in the length of hospitalization and mortality.

Identifying these patients at risk is essential to limit complications (pneumonia, reintubation, inadequate refeeding, etc.). The benchmark test to objectify vocal cord palsy is to perform a nasofibroscopy requiring equipment and the intervention of an ENT doctor or thoracic surgeon.

A physiotherapist can also perform a preliminary swallowing test by evaluating several criteria.

The aim of this study is to compare the concordance of results between nasofibroscopy and that by preliminary swallowing test, two procedures performed in the screening of vocal cord paralysis in a surgical intensive care unit and a thoracic surgery ward.

Patients will be included before the surgery. During this inclusion visit, we will perform a preoperative swallowing test.

Immediately after surgery (H2-H24 after extubation), we will perform a preliminary swallowing test, an ultrasound examination of the vocal cords and a nasofibroscopy to determine the mobility of the vocal cords. A physiotherapist will carry out the first two assessments. An ENT physician will perform the nasofibroscopy. The ENT physician performing the nasofibroscopy will not know the conclusions of the tests carried out by the physiotherapist immediately after the operation.

At last, on day 4 after extubation, we will repeat the preliminary swallowing test and the ultrasound examination to measure the evolution of cord mobility.

Initial evaluation and secondary evaluation (day 4) will be performed by two different physiotherapists in order to allow blinding between the two stages of the procedure.

45 days after the surgery, we will realize a follow-up on medical file and mark the end of the research.

We want to include 72 patients over an 18 months period.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old)
* Patient who is scheduled for a major left lung resection surgery (segmentectomy, lobectomy, pneumonectomy) or a right lung resection with upper lymph node dissection in the context of lung cancer
* Patient who capable to read and understand the patient information and consent.
* Patient capable to read and sign the consent form
* Patient with social insurance
* Woman of childbearing age with effective contraception (see WHO definition), postmenopausal woman (≥ 12 months of amenorrhea not induced by therapy)
* Negative urine pregnancy test

Exclusion Criteria:

* History of swallowing or eating disorders,
* Neurological history with known sequelae or cognitive disorders
* Preoperative nasogastric tube feeding
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection, under guardianship or curatorship,
* Pregnant or breastfeeding woman
* Patient participating in another clinical trial with the same primary outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
discreapancies between preliminary swallowing test and nasofibroscopy | 2 hours after extubation to 24 hours after extubation
  the number of discrepancies between the two test, namely the times when the two tests do not reach the same conclusion after the patients's extubation

SECONDARY OUTCOMES:
Prevalence of swallowing disorders pre-existing to planned surgery, | inclusion
  established according to the results of the swallowing test carried out by a physiotherapist
performance of the preliminary swallowing test | 2 hours after extubation to 24 hours after extubation
  * Sensitivity: The number of patients for whom the two tests reach the same conclusion among those with disorders according to the nasofibroscopy test
  * Specificity: The number of patients for whom the two tests reach the same conclusion among those who have no disorder according to the nasofibroscopy test
Performance of the ultrasound examination | 2 hours after extubation to 24 hours after extubation
  * Sensitivity: The number of patients for whom the two tests reach the same conclusion among those with disorders according to the nasofibroscopy test
  * Specificity: The number of patients for whom the two tests reach the same conclusion among those who have no disorder according to the nasofibroscopy test
- Proportion of patients for whom the score of the preliminary swallowing test on day 4 is different than that obtained for the same test carried out immediately postoperatively | Between (2 hours after extubation to 24 hours after extubation) and Day 4
  - Proportion of patients for whom the score of the preliminary swallowing test on day 4 is different than that obtained for the same test carried out immediately postoperatively
Proportion of patients for whom the score of the ultrasound examination of the vocal cords on day 4 is different than that obtained for the same test carried out immediately postoperatively | Between (2 hours after extubation to 24 hours after extubation) and Day 4
  Proportion of patients for whom the score of the ultrasound examination of the vocal cords on day 4 is different than that obtained for the same test carried out immediately postoperatively
Assessment of the discomfort felt during the 3 tests | 2 hours after extubation to 24 hours after extubation
  Assessment of the discomfort felt during the 3 tests carried out using a numerical scale from 0 to 10
Prevalence of postoperative complications according to the grade of the Clavien-Dindo classification | 30 days after surgery
  Prevalence of postoperative complications according to the grade of the Clavien-Dindo classification (within 30 days after surgery). The national database EpiThor provides this information.

CONTACTS AND LOCATIONS:
Overall Officials: Baptiste MICHAUX, physiotherapist, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No